CLINICAL TRIAL: NCT02259426
Title: A Double Blind Randomized Controlled Trial of Dihydroartemisinin-piperaquine Alone and in Combination With Single Dose Primaquine to Reduce Post-treatment Malaria Transmission.
Brief Title: Dihydroartemisinin-piperaquine With Low Dose Primaquine to Reduce Malaria Transmission
Acronym: DAPPI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Radboud University Medical Center (Other); International Centre of Insect Physiology and Ecology (ICIPE) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAPPI-1
Record Dates: First submitted 2014-09-29; First posted 2014-10-08 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Malaria; Asymptomatic Malaria; Plasmodium Falciparum
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Primaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dihydroartemisínin-piperaquine (Artekin) (Active Comparator): Dihydroartemisínin-piperaquine combination alone
  Interventions: Drug: Dihydroartemisinin-piperaquine combination (Artekin)
- Dihydroartemisinin-piperaquine, Primaquine (Experimental): Dihydroartemisinin-piperaquine with single-dose 0.25mg/kg Primaquine
  Interventions: Drug: Dihydroartemisinin-piperaquine combination (Artekin); Drug: Primaquine

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine combination (Artekin)
Drug: Primaquine — Single-dose 0.25mg/kg
  Arms: Dihydroartemisinin-piperaquine, Primaquine

SUMMARY:
Primaquine (PQ) is currently the only available drug that can clear the mature transmission stages of P. falciparum parasites. PQ was previously shown to clear gametocytes that persist after artemisinin-combination therapy. A major caveat to the use of primaquine in mass adminsitrations for the reduction of malaria transmission is that metabolism of the drug in individuals with glucose-6 phosphate dehydrogenase (G6PD) deficiency can lead to transient haemolysis. The haemolytic side effect of PQ is dose-related. Haemolysis is more commonly observed after prolonged PQ treatment but has also been observed in African populations following a single dose of PQ. This haemolysis was self-limiting, largely restricted to G6PD deficient individuals and did not lead to clinical symptoms. Nevertheless, any drug-induced haemolysis is reason for concern and the World Health Organization has therefore reduced the recommended dose of single low dose primaquine from 0.75mg/kg to 0.25mg/kg. This dosage is deemed safe without prior G6PD or Hb screening. However, there is limited direct evidence on the extent to which this dosage of PQ prevents malaria transmission to mosquitoes.

In the current study, the investigators will assess the efficacy of DP in combination with low-dose PQ to prevent onward malaria transmission. The investigators will perform the investigators study in individuals aged 5-15 years who are carry microscopically detectable densities of P. falciparum gametocytes. This age group is chosen because asexual parasite carriage and gametocyte carriage are common in this age group. All enrolled individuals will receive a full three-day course of DP, and will be randomized to receive a dose of primaquine or placebo with their third dose. Efficacy will be determined based on gametocyte carriage during follow-up, measured by molecular methods. For all individuals, the effect of treatment on infectivity to mosquitoes will be assessed by membrane feeding assays at two time points.

ELIGIBILITY:
Inclusion Criteria:

* Microscopically detectable P. falciparum gametocyte carriage

Exclusion Criteria:

* Age < 5 years or > 15 years
* Non-falciparum malaria co-infection
* Malaria parasite density ≥ 200,000 parasites/µL
* Clinical symptoms indicating severe malaria
* Axillary temperature ≥ 39°C
* Body Mass Index (BMI) below 16 or above 32 kg/m2
* Haemoglobin concentration below 9.5 g/dL
* Anti-malarials taken in last 2 days
* For women: Pregnancy (assessed by clinical examination and urine pregnancy test) or lactation
* Known hypersensitivity to DP or PQ
* History and/or symptoms indicating chronic illness
* Current use of tuberculosis or anti-retroviral medication
* Unable to give written informed consent
* Unwillingness to participate in two membrane feeding assays
* Travel history to Angola, Cameroon, Chad, Central African Republic, Congo, DR Congo, - Equatorial Guinea, Ethiopia, Gabon, Nigeria and Sudan
* Family history of congenital prolongation of the QTc interval or sudden death or with any other clinical condition known to prolong the QTc interval such as history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease
* Taking drugs that are known to influence cardiac function and to prolong QTc interval, such as class IA and III: neuroleptics, antidepressant agents, certain antibiotics including some agents of the following classes - macrolides, fluoroquinolones, imidazole, and triazole antifungal agents, certain non-sedating antihistaminics (terfenadine, astemizole) and cisapride
* Known disturbances of electrolyte balance, e.g. hypokalaemia or hypomagnesaemia
* Taking drugs which may be metabolized by cytochrome enzyme CYP2D6 (e.g., flecainide, metoprolol, imipramine, amitriptyline, clomipramine)
* Blood transfusion within last 90 days

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Gametocyte prevalence on day 7 after initiation of treatment | day 7 of follow-up
  Gametocyte prevalence on day 7 after initiation of treatment is measured by molecular methods.

SECONDARY OUTCOMES:
Transmission to Anopheles gambiae mosquitoes | Day 3 and 7 during follow-up
  Mosquito membrane feeding assays will be used to determine the proportion of infected mosquitoes and the oocyst burden in infected mosquitoes.
Haematological recovery | 14 days during follow-up
  Haemoglobin concentration will be determined at enrolment and on days 2, 3, 7 and 14 during follow-up. Haemoglobin concentration will be presented as grams per decilitre and as concentration relative to enrollment value.
Gametocyte sex-ratio | 14 days of follow-up
  The ratio of male:female gametocytes will be determined at enrolment and on days 2, 3, 7 and 14 during follow-up by qRT-PCR.
Gametocyte carriage during follow-up | 14 days during follow-up
  Gametocyte prevalence at enrolment and on days 2, 3, 7 (primary outcome measure), and 14 during follow-up. The duration of gametocyte carriage in days will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Teun Bousema, PhD, Principal Investigator — Radboud university medical center, London School of hygiene and tropical medicine; Patrick Sawa, MD, Principal Investigator — ICIPE
Locations (1):
- ICIPE, Mbita, Nyanza, Kenya